CLINICAL TRIAL: NCT06048640
Title: Effects of Dynamine Ingestion on Various Indices of Sustained Energy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: #CSI-08-2022-001
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Energy
MeSH Terms: interventions — methylliberine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 100 mg of placebo (cellulose)
  Interventions: Dietary Supplement: Dynamine (methylliberine)
- Active (Active Comparator): 100 mg of Dynamine (methylliberine)
  Interventions: Dietary Supplement: Dynamine (methylliberine)

INTERVENTIONS:
Dietary Supplement: Dynamine (methylliberine) — Dynamine (methylliberine) is a purine alkaloid found in the kucha leaf, and available to consumers as a dietary supplement.

SUMMARY:
This study is a randomized, placebo-controlled, double-blind, within-subject crossover trial of 25 men and women. The objective of this study is to assess the effects of Dynamine (methylliberine) supplementation on overall well-being including energy, sustained energy, mental stamina, focus, concentration, motivation to accomplish difficult tasks, drive, vigor, positive outlook, maintaining a healthy mood, feelings of well-being, and resilience to stress.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blind, within-subject crossover trial of 25 men and women. Dynamine (methylliberine) is a caffeine metabolite and purine alkaloid found in the kucha tea leaf. Dynamine has become a popular dietary supplement with consumers due to its neuro-energetic effects. Previous research has shown Dynamine can improve energy, mood and focus without the cardiovascular effects of elevating heart rate or blood pressure.

In this study, participants will attend 5 study visits. During Visit 1, participants will be screened for participation (i.e., medical history, routine blood work, background baseline diet). During Visits 2 and 4, participants will complete baseline testing including subjective questionnaires that assess energy, sustained energy, mental stamina, focus, concentration, motivation to accomplish difficult tasks, drive, vigor, positive outlook, maintaining a healthy mood, feelings of well-being, resilience to stress in addition to completion of a series of an objective neuropsychological test (Stroop test) to assess mental processing, cognitive flexibility, and attention. After three-4- days of supplementation, participants will return for Visit 3 and 5 where they will take a 4th dose of Dynamine or placebo and repeat the testing outlined at previous baseline visits.

ELIGIBILITY:
Inclusion Criteria:

* provide voluntary signed and dated informed consent
* in good health as determined by physical examination and medical history
* between the ages of 21 and 55 years
* body mass index (BMI) of 18.5-27 kg•m-2
* agrees to abstain from exercise and alcohol for 24 hours prior to each study visit
* agrees to abstain from coffee and caffeinated beverages for 12 hours prior to each study visit
* normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg
* normal seated, resting heart rate (<90 per minute)
* willing to duplicate their previous 24-hour and fast for 8 hours prior each study visit

Exclusion Criteria:

* a history of diabetes or pre-diabetes
* a history of malignancy in the previous 5 years except for non-melanoma skin cancer
* prior gastrointestinal bypass surgery
* known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism
* any chronic inflammatory condition or disease
* a known allergy to any of the ingredients in the supplement or the placebo
* currently participating in another research study with an investigational product or have been in another research study in the previous 30 days
* a caffeine intake of three or more cups of coffee or equivalent (>400 mg) per day
* uses corticosteroids or testosterone replacement therapy (ingestion, injection, or transdermal)
* had any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the participant at increased risk of harm if they were to participate

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Concentration | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Concentration as measured by a 10 cm visual analogue scale, where higher values represent better concentration.
Motivation | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Motivation as measured by a 10 cm visual analogue scale, where higher values represent greater motivation.
Mood | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Mood as measured by a 10 cm visual analogue scale, where higher values represent better mood.
Energy | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Energy as measured by a 10 cm visual analogue scale, where higher values represent increased energy.
Sustained Energy | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Sustained energy as measured by a 10 cm visual analogue scale, where higher values represent increased sustained energy.
Well-being | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Well-being as measured by a 10 cm visual analogue scale, where higher values represent improved feelings of well-being.
Cognitive function | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Cognitive function as measured by the Stroop Test.
Cognitive flexibility | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Cognitive flexibility as measured by the Trail Making Test.

SECONDARY OUTCOMES:
Systolic blood pressure | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Systolic blood pressure in mm of mercury.
Diastolic blood pressure | Change from baseline to 60 minutes, 120 minutes, and 180 minutes post-baseline.
  Diastolic blood pressure in mm of mercury.

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Raub, RN, BSN, Principal Investigator — The Center for Applied Health Sciences
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided